CLINICAL TRIAL: NCT00015951
Title: A Phase II Study of the Recombinant Human Monoclonal Anti-Vascular Endothelial Growth Factor Antibody (rhuMAB VEGF) Bevacizumab (NSC #704865, IND # 7,921) Administered in Times Sequential Combination With Cytosine Arabinoside (Ara-C) and Mitoxantrone for Adults With Refractory and Relapsed Acute Myelogenous Leukemias (AMLs)
Brief Title: Bevacizumab, Cytarabine, and Mitoxantrone on Treating Patients With Hematologic Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Maryland Greenebaum Cancer Center (Other)
Responsible Party: UM Greenebaum Cancer Center
Purpose: Treatment
Other Study IDs: CDR0000068576; MSGCC-0076; NCI-2490
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: recurrent adult acute myeloid leukemia; relapsing chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; secondary acute myeloid leukemia; previously treated myelodysplastic syndromes; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Blast Crisis; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — Bevacizumab; Cytarabine; Mitoxantrone

INTERVENTIONS:
Biological: bevacizumab
Drug: cytarabine
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Monoclonal antibodies such as bevacizumab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Combining monoclonal antibody therapy with chemotherapy may be an effective treatment for hematologic cancer.

PURPOSE: Phase II trial to study the effectiveness of bevacizumab combined with cytarabine and mitoxantrone in treating patients who have hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical effectiveness of bevacizumab, cytarabine, and mitoxantrone in patients with poor-risk hematologic malignancies.
* Determine the toxic effects of this regimen in these patients.
* Determine whether this regimen can induce cell apoptosis in these patients.
* Determine the effects of bevacizumab on coagulation profiles in these patients.

OUTLINE: This is a multicenter study.

Patients receive cytarabine IV continuously over 72 hours on days 1-3, mitoxantrone IV over 30-60 minutes on day 4, and bevacizumab IV over 90 minutes on day 8 in the absence of disease progression or unacceptable toxicity. Patients achieving partial or complete remission may receive a second course of therapy beginning approximately 30 days after the completion of the first course.

Patients are followed until death.

PROJECTED ACCRUAL: A total of 12-45 patients will be accrued for this study within 1-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed poor-risk hematologic malignancy

  * Relapsed or refractory acute myelogenous leukemia (AML)

    * Primary induction failure
    * Myelodysplasia(MDS)-related AML
    * Secondary AML
  * Relapsed or refractory MDS

    * Primary induction failure
    * Refractory anemia with excess blasts (RAEB)
    * RAEB in transformation
    * Chronic myelomonocytic leukemia
  * Chronic myelogenous leukemia in blast crisis
* Failure of prior primary induction therapy or relapse after achieving complete remission allowed only if no more than 3 courses of prior induction/reinduction therapy were received
* No hyperleukocytosis (50,000 or more leukemic blasts/mm3)
* No active CNS leukemia

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics
* No disseminated intravascular coagulation

Hepatic:

* AST/ALT no greater than 2 times normal
* Alkaline phosphatase no greater than 2 times normal
* Bilirubin no greater than 1.5 times normal

Renal:

* Creatinine no greater than 1.5 times normal

Cardiovascular:

* LVEF at least 45% by MUGA or echocardiogram
* No myocardial infarction within the past 3 months
* No history of severe coronary artery disease
* No cardiomyopathy
* No New York Heart Association class III or IV heart disease (congestive heart failure)

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active uncontrolled infection
* No history of cytarabine-related neurotoxicity
* No evidence of graft-versus-host disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 week since prior hematopoietic growth factors including epoetin alfa, filgrastim (G-CSF), and sargramostim (GM-CSF)
* At least 1 week since prior interleukin-3 or interleukin-11
* At least 4 weeks since prior autologous stem cell transplantation
* At least 90 days since prior allogeneic stem cell transplantation
* No other concurrent immunotherapy

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy and recovered
* No prior cytarabine administered as a 72-hour continuous infusion followed by mitoxantrone IV over 30 minutes
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* At least 2 weeks since prior immunosuppressive therapy
* No other concurrent investigational or commercially available antitumor therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04; Primary Completion 2003-04 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith E. Karp, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (3):
- United States (3):
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland